CLINICAL TRIAL: NCT01845012
Title: Evaluation of Daily HemoDialysis at Low Dialysate Flow in Patients Previously Treated With Conventional Hemodialysis
Acronym: HDQ200
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been prematurely halted because of failure of patient recruitment.
Sponsor: Association Pour L'utilisation Rein Artificiel Région Lyonnaise (Other)
Collaborators: Association Nationale pour la promotion de la Dialyse Quotidienne (ANDIQ, France) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A00307-36
Record Dates: First submitted 2013-04-11; First posted 2013-05-03 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: End Stage Renal Disease
Keywords: Short daily hemodialysis; Low dialysate flow; End stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily hemodialysis at low dialysate flow (Experimental)
  Interventions: Other: Daily hemodialysis at low dialysate flow

INTERVENTIONS:
Other: Daily hemodialysis at low dialysate flow — Daily hemodialysis at low dialysate flow during 3 months: 6 times 2h to 2h30 per week at a dialysate flow rate of 200 ml/min in order that the total duration of weekly dialysis is equivalent to the duration of weekly dialysis during the last 3 months of conventional hemodialysis. Other parameters of dialysis (dialysate, dialysis machine, generator, blood flow, anticoagulation) are the same as the reference period of conventional hemodialysis.

SUMMARY:
HDQ 200 is an interventional multicenter study. This is a before-and-after design in which the patient is his own control. The main objective of the study is to determine the percentage of success of a procedure of daily hemodialysis at low dialysate flow. All patients treated with conventional hemodialysis, for at least 3 months and clinically stable, can be included in the study. Their 3 months data prior to inclusion is collected retrospectively. These 3 months of conventional hemodialysis are the reference period. Patients are then treated with daily hemodialysis at low dialysate flow for 3 months. During this 3 months period, the same data as during the period of conventional hemodialysis are collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who give voluntary signed informed consent
* Patients affiliated with the French universal health care system or similar
* For women of childbearing potential: serum or urine negative pregnancy test
* Patients treated with conventional hemodialysis (3 times 4h to 5h per week at at least a dialysate flow rate of 500 ml/min) for at least 3 months and clinically stable (investigator assessment)
* Bipuncture patients (or with double lumen central venous catheter) with stable vascular access and easy to puncture
* Patients willing to be treated with daily hemodialysis at low dialysate flow during the study period (6 times 2h to 2h30 per week at a dialysate flow rate of 200 ml/min in order that the total duration of weekly dialysis is equivalent to the duration of weekly dialysis during the last 3 months of conventional hemodialysis)

Exclusion Criteria:

* Pregnant women or women who could become pregnant during the study (planned pregnancy within 3 months)
* Patients not affiliated with the French universal health care system
* Minor patients
* Patients who are protected adults according to the terms of the law (French public health laws).
* Refusal to give consent
* Patients simultaneously participating in another trial that may interfere with the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients for whom the period of daily hemodialysis at low dialysate flow will be a success. | Every 2 weeks during 3 months.
  Definition of success: if during the period of daily hemodialysis at low dialysate flow, the patient maintains the absolute value of their pre-dialysis serum creatinine (mid-week dialysis) below the upper limit of the confidence interval established during the 3 months prior to inclusion on 7 values: measurements every 2 weeks for 3 months (retrospective data) and inclusion measurement included (Day 0).
  Daily hemodialysis at low dialysate flow will be considered as a failure if pre-dialysis serum creatinine values exceed twice successively the upper limit of the confidence interval established for the patient.

SECONDARY OUTCOMES:
Number of patients who stopped the daily hemodialysis at low dialysate flow (patient or investigator's decision). | 3 months.
Number of patients who maintained a satisfactory clinical condition (investigator assessment) during the period of daily hemodialysis at low dialysate flow. | 3 months.
Evaluation of weight. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): every 2 weeks.
Evaluation of blood pressure. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): every 2 weeks.
Evaluation of heart rate. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): every 2 weeks.
Evaluation of body mass index. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): every 2 weeks.
Evaluation of metabolic parameters. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): every 2 weeks.
Evaluation of hematological parameters. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): every 2 weeks.
Evaluation of inflammation parameters. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): monthly.
Evaluation of nutrition parameters. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): monthly.
Evaluation of iron parameters. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): monthly.
Change in hormones. | At inclusion and at 3 months.
  Measurement at inclusion represent the retrospective period of 3 months in conventional hemodialysis. Measurement at 3 months represent the prospective period of 3 months in daily hemodialysis at low dialysate flow.
Composite measurement of treatments. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): at each hemodialysis.
  A listing of all the therapeutics changes made between the two dialysis periods will be provided (e.g. dose of erythropoietin, phosphate binders, antihypertensive drugs, other treatments)
Composite measurement of technical dialysis parameters. | During 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
  Detail of time frame during 3 months (retrospectively and prospectively): every 2 weeks.
  A listing of all the technical dialysis changes made between the two dialysis periods will be provided (e.g. urea clearance of the dialysis machine, effective duration of dialysis, ultrafiltration time rate and per dialysis, type of access, blood flow, dialysate flow rate, dialysate composition and anticoagulation method).
List of symptoms and incidents between two hemodialysis, evaluation of hemodialysis tolerance, clinical assessment of the vascular access and possible local complications. | At each hemodialysis during 3 months (retrospectively and prospectively).
  The retrospective study period is 3 months of conventional hemodialysis. The prospective study period is 3 months of daily hemodialysis at low dialysate flow.
Change in quality of life. | At inclusion and at 3 months.
  Measurement at inclusion represent the retrospective period of 3 months in conventional hemodialysis. Measurement at 3 months represent the prospective period of 3 months in daily hemodialysis at low dialysate flow.
Change in pain. | At inclusion and at 3 months.
  Measurement at inclusion represent the retrospective period of 3 months in conventional hemodialysis. Measurement at 3 months represent the prospective period of 3 months in daily hemodialysis at low dialysate flow.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Laville, MD, PHD, Principal Investigator — Hospices Civils de Lyon, Centre Hospitalier Lyon Sud, Service de Néphrologie Bâtiment 3C, 3ème étage, Chemin du grand Revoyet 69495 PIERRE-BENITE
Locations (13):
- Cliniques universitaires St Luc, Brussels, Belgium
- France (12):
  - ECHO Angers, Angers
  - CTMR Saint Augustin, Bordeaux
  - CHPC, Cherbourg
  - CHU Grenoble, Grenoble
  - ANIDER, Le Petit-Quevilly
  - AURAL, Lyon
  - Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon
  - AGDUC Meylan, Meylan
  - AURA - Paris, Paris
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - ECHO Nantes, Rezé
  - Centre Hospitalier de Vichy, Vichy